CLINICAL TRIAL: NCT02737449
Title: CorEvitas Japan Rheumatoid Arthritis (RA) Registry
Status: Active, not recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-RA-102
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to prospectively study the comparative effectiveness and comparative safety of approved therapies for RA in a Japanese cohort of patients treated by rheumatologists. This includes assessing the incidence of adverse events of special interest, in a real-world population of rheumatoid arthritis patients. Secondary objectives include analyzing the epidemiology and natural history of the disease, comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
The design is a prospective, multicenter, non-interventional, observational study for patients with RA who are newly prescribed eligible medications at the time of enrollment into the registry. The drug is prescribed per the physician's decision which precedes the decision to enroll the patient into the registry. Longitudinal follow-up data is obtained via CorEvitas Questionnaires completed by both patients and their treating rheumatologists during routine clinical practice. The Enrollment and Follow-Up Questionnaires capture data on patient demographics, targeted medical history including a history of all prior treatments for RA, smoking history, disease duration, disease severity, disease activity, laboratory results, comorbidities, hospitalizations and other targeted safety events.

The study will also monitor a range of clinical effectiveness, patient reported outcomes (PROs), health economic, and safety outcomes, including infections, malignancies and cardiovascular events, among other safety outcomes. Standard components of the European League Against Rheumatism (EULAR) (Disease Activity Score -28 joint count) and American College of Rheumatology (ACR) response criteria, including tender and swollen 28 joint counts, physician and patient global assessment, morning stiffness and pain will be collected at all study visits to enable comparisons of composite disease activity scores (e.g. remission) and response criteria. disease activity score (DAS)-28 erythrocyte sedimentation rates (ESR) will be calculated where possible, as Japanese physicians routinely collect ESR on a more regular basis than U.S. physicians. Composite indices of disease activity, clinical disease activity index (CDAI), DAS, and ACR scores may be calculated from the elements in the CorEvitas Questionnaire for publication. In addition, PROs will be collected via instruments including the EuroQol (EQ)-5D, health assessment questionnaire (HAQ)-DI, and work productivity activity impairment instrument (WPAI) questionnaire.

A primary objective of the registry is analysis of comparative safety. The registry may be linked to other registries for the purposes including comparative safety or outcome studies. The program-specific subject identifier number (ID) will be collected for subjects that participate or have participated in a post-market surveillance study. The ID will be used for to ensure the accuracy of safety reporting to regulators by reducing duplicate reports Note that this study has not been submitted to a United States institutional review board. It has been approved by Japanese Authorities.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be diagnosed with rheumatoid arthritis according to the 1987 ACR or the ACR/EULAR 2010 Rheumatoid Arthritis Classification Criteria
* The subject must be at least 18 years of age or older
* The subject must be able and willing to provide written consent
* The subject must be prescribed or switching to an eligible medication for the first time ever at the Enrollment Visit. History of concomitant treatment with other eligible medications does not exclude a subject from enrollment.

Exclusion Criteria:

* The subject is unable or unwilling to provide informed consent to participate in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CorEvitas Japan RA Registry has a target enrollment of approximately 2,600 subjects with no defined upper limit on enrollment.This study will recruit patients from approximately 60 clinical sites from a broad geographic distribution in Japan; however, there is no defined upper or lower limit on the number of sites expected to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-07; Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of adverse events (AEs) will be measured. | e outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
  Number of patients who develop malignancy, cardiovascular disease, serious infection, inflammatory bowel syndrome, hepatic events, neurological events and general serious adverse events (SAEs) in Japanese clinical practice will be assessed in subjects receiving Conventional synthetic DMARDs, JAK inhibitors, Anti-TNF biologic DMARDs, and Non-TNF biologic DMARDs as standard of care.

SECONDARY OUTCOMES:
The number of tender and swollen joints, 28 joint counts, will be recorded as a measure of disease activity. | 1. the outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Patient pain assessment will be collected using visual analogue scale measurements (VAS) | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Physician global disease severity assessment will be collected using VAS | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Patient global disease severity assessment will be collected using VAS. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
The duration of morning stiffness will be recorded in minutes or hours. enrollment and subsequent visits | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
The severity of morning stiffness, stiffness and associated pain, will be recorded using VAS. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
DAS-28 ESR rates will be calculated. . | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Composite indices of disease activity: CDAI score, will be calculated from the elements in the CorEvitas Questionnaires. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Composite indices of disease activity, ACR score, will be calculated from the elements in the CorEvitas Questionnaires. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
Composite indices of disease activity, DAS score, will be calculated from the elements in the CorEvitas Questionnaires. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
PROs will be collected via instruments including the EQ-5D questionnaire. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
PROs will be collected via instruments including the HAQ-DI questionnaire. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.
PROs will be collected via instruments including the WPAI questionnaire. | The outcome measure will be assessed at enrollment and at each subsequent study visit, approximately every 6 months, through study completion, an average of 8 years.

IPD SHARING:
Plan to Share IPD: No